CLINICAL TRIAL: NCT00671307
Title: Phase 1b Randomized, Double-blind, Placebo-controlled, Ascending Single Dose Infusion Trial of the Pharmacokinetics of Rhu-pGelsolin in Patients With Decreased Natural Gelsolin Levels
Brief Title: Ascending Single Dose Study of Rhu-pGelsolin in Patients With Decreased Gelsolin Levels
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Critical Biologics Corporation (Industry)
Responsible Party: Richard Straube, MD/ Chief Medical Officer, Critical Biologics Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBC101
Record Dates: First submitted 2008-04-30; First posted 2008-05-05 (Estimated); Last update posted 2010-09-29 (Estimated); Status verified 2010-04

CONDITIONS: Low Gelsolin; Trauma; Infection; Burns
Keywords: Gelsolin; Trauma; Pneumonia; Peritonitis; Burn; Infection; Sepsis; Systemic Inflammatory Response Syndrome
MeSH Terms: conditions — Wounds and Injuries; Infections; Burns; Meretoja syndrome; Pneumonia; Peritonitis; Sepsis; Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Low dose (Experimental): 3 mg/kg of rhu-pGelsolin given as an IV infusion over 1 hour
  Interventions: Drug: rhu-pGelsolin
- Mid-dose (Experimental): 6 mg/kg of rhu-pGelsolin given as an IV infusion over 1 hour
  Interventions: Drug: rhu-pGelsolin
- High dose (Experimental): 6 mg/kg of rhu-pGelsolin given a an IV infusion over 1 hour once a day for 3 days
  Interventions: Drug: rhu-pGelsolin

INTERVENTIONS:
Drug: rhu-pGelsolin — IV formulation of recombinant plasma gelsolin formulated as 10 mg/ml given as a single IV infusion over 1 hour
  Other Names: Recombinant plasma gelsolin; CBC-100; Solinex
  Arms: High dose; Low dose; Mid-dose
Drug: Placebo — Vehicle control given as IV infusion over 1 hour
  Other Names: Vehicle control
  Arms: Placebo

SUMMARY:
This study is designed to assess the pharmacokinetics and safety of an infusion of a single dose of recombinant plasma gelsolin (rhu-pGelsolin) when given to patients admitted to the Intensive Care Unit with documented low levels of natural gelsolin. It is believed that this drug will raise the gelsolin levels in these patients and decrease the probability that they will develop complications from their underlying disease such as organ system failure or death.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, ascending single dose of rhu-pGelsolin infusion study. Thirteen subjects (10 active and 3 placebo) will be dosed at 3 mg/kg and 5 subjects (3 active and 2 placebo) will be dosed at 6 mg/kg. In addition, twenty-two subjects (18 active and 4 placebo) will be dosed at 6 mg/kg per day for 3 days. The Data Safety Monitoring Committee (DSMC) and Steering Committee will review the preceding dose safety data, and agree the tolerability prior to the enrolment for next higher dose. Blood samples will be collected during 1 hour infusion through 72 hours post dose for PK assessment after each dose.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Documented gelsolin level <100 mg/mL
* Admission to ICU
* Women of child-bearing age have a negative pregnancy test
* Multiple Organ Failure score < 4
* Catheter present through which blood samples can be taken
* Written Informed Consent obtained

Exclusion Criteria:

* Participation in other investigational treatment protocols
* Patients <18 years of age
* Patients who have a modified Multiple Organ Failure score of >=4
* Patient, who in the opinion of the Principal Investigator, are unlikely to be in the ICU for >48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-03; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of plasma gelsolin | 72 hours

SECONDARY OUTCOMES:
Adverse events and the development of anti-rhu-pGelsolin antibodies | 3 months
Pharmacodynamics of sepsis biomarkers | 72 hours
Clinical outcomes (mortality, duration of ICU stay, duration of ventilator support, duration of hospital stay) | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Wai M Chan, MBBS, Principal Investigator — Queen Mary Hospital, Hong Kong; Selene Tam, PhD, Study Director — University of Hong Kong; Clinical Trials Centre; Richard C Straube, MD, Study Chair — Critical Biologics Corporation
Locations (1):
- Queen Mary Hospital; University of Hong Kong, Hong Kong, SAR, Hong Kong

REFERENCES:
- [Background] Lee PS, Waxman AB, Cotich KL, Chung SW, Perrella MA, Stossel TP. Plasma gelsolin is a marker and therapeutic agent in animal sepsis. Crit Care Med. 2007 Mar;35(3):849-55. doi: 10.1097/01.CCM.0000253815.26311.24. PMID 17205019
- [Background] Lee PS, Drager LR, Stossel TP, Moore FD, Rogers SO. Relationship of plasma gelsolin levels to outcomes in critically ill surgical patients. Ann Surg. 2006 Mar;243(3):399-403. doi: 10.1097/01.sla.0000201798.77133.55. PMID 16495706
- [Background] Christofidou-Solomidou M, Scherpereel A, Solomides CC, Christie JD, Stossel TP, Goelz S, DiNubile MJ. Recombinant plasma gelsolin diminishes the acute inflammatory response to hyperoxia in mice. J Investig Med. 2002 Jan;50(1):54-60. doi: 10.2310/6650.2002.33518. PMID 11813829
- [Background] Rothenbach PA, Dahl B, Schwartz JJ, O'Keefe GE, Yamamoto M, Lee WM, Horton JW, Yin HL, Turnage RH. Recombinant plasma gelsolin infusion attenuates burn-induced pulmonary microvascular dysfunction. J Appl Physiol (1985). 2004 Jan;96(1):25-31. doi: 10.1152/japplphysiol.01074.2002. Epub 2003 May 2. PMID 12730154
- [Background] Mounzer KC, Moncure M, Smith YR, Dinubile MJ. Relationship of admission plasma gelsolin levels to clinical outcomes in patients after major trauma. Am J Respir Crit Care Med. 1999 Nov;160(5 Pt 1):1673-81. doi: 10.1164/ajrccm.160.5.9807137. PMID 10556139
- [Background] DiNubile MJ, Stossel TP, Ljunghusen OC, Ferrara JL, Antin JH. Prognostic implications of declining plasma gelsolin levels after allogeneic stem cell transplantation. Blood. 2002 Dec 15;100(13):4367-71. doi: 10.1182/blood-2002-06-1672. Epub 2002 Aug 1. PMID 12393536
- [Background] Suhler E, Lin W, Yin HL, Lee WM. Decreased plasma gelsolin concentrations in acute liver failure, myocardial infarction, septic shock, and myonecrosis. Crit Care Med. 1997 Apr;25(4):594-8. doi: 10.1097/00003246-199704000-00007. PMID 9142022